CLINICAL TRIAL: NCT00303563
Title: A Randomized, Double-blind Study to Compare the Effect of RO4402257 Monotherapy and Methotrexate Monotherapy on Disease Response in Patients With Active Rheumatoid Arthritis.
Brief Title: A Study of P38 Inhibitor (4) Monotherapy in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA18604
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: P38 Inhibitor (4)
- 2 (Experimental)
  Interventions: Drug: P38 Inhibitor (4)
- 3 (Experimental)
  Interventions: Drug: P38 Inhibitor (4)
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: P38 Inhibitor (4) — 50mg po qd
  Arms: 1
Drug: P38 Inhibitor (4) — 150mg po qd
  Arms: 2
Drug: P38 Inhibitor (4) — 300mg po qd
  Arms: 3
Drug: Placebo — po qd
  Arms: 4

SUMMARY:
This 4 arm study will compare the safety and efficacy, with regard to reduction of signs and symptoms, of P38 Inhibitor (4) (50, 150 or 300mg po qd) monotherapy versus methotrexate monotherapy in adult patients with active rheumatoid arthritis. Patients will be randomized to receive one of 3 doses of P38 Inhibitor (4) or methotrexate. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >18 years of age, with active RA;
* receiving treatment for RA on an outpatient basis;
* females of child-bearing potential, or nonsterilized males with partners of child-bearing potential, must use reliable contraception during, and for 4 weeks after, the study.

Exclusion Criteria:

* major surgery within 8 weeks prior to screening;
* rheumatic autoimmune disease or inflammatory joint disease other than RA;
* treatment with methotrexate within 8 weeks of baseline;
* concurrent use of DMARDs, including anti-TNF or other biologic therapy for RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | Week 12

SECONDARY OUTCOMES:
Percentage of patients with ACR 50/70 response. | Week 12
Change in ACR core set, DAS 28, FACIT-F fatigue assessment, AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- United States (21):
  - Anniston, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Escondido, California
  - Loma Linda, California
  - Stamford, Connecticut
  - Morton Grove, Illinois
  - South Bend, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Belmont, North Carolina
  - Bend, Oregon
  - Danville, Pennsylvania
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
- Canada (4):
  - Edmonton, Alberta
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Toronto, Ontario
- Croatia (2):
  - Rijeka
  - Split
- Czechia (4):
  - České Budějovice
  - Prague
  - Terezín
  - Zlín
- France (5):
  - Brest
  - Corbeil-Essonnes
  - Montpellier
  - Paris
  - Rouen
- Italy (4):
  - Brescia
  - Genova
  - Pavia
  - Roma
- Mexico (2):
  - Guadalajara
  - Miexico City
- Romania (2):
  - Brasov
  - Bucharest
- Belgrade, Serbia
- South Africa (3):
  - Bloemfontein
  - Johannesburg
  - Pretoria
- Spain (8):
  - A Coruña
  - Barcelona
  - Granada
  - Jerez de la Frontera
  - Madrid
  - Oviedo
  - Palma de Mallorca
  - Seville
- Taiwan (3):
  - Kaohsiung City
  - Taoyuan District
  - Tapei